CLINICAL TRIAL: NCT02900599
Title: Predicting Treatment and Care Difficulties Among HIV Infected Patients
Acronym: PREDIVI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: PREDIVI
Record Dates: First submitted 2016-09-06; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: HIV
Keywords: HIV; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observationnal (no intervention)

SUMMARY:
Much of HIV is related to behaviour: sexual risk taking, late diagnosis, adherence to antiretroviral therapy, follow up, disclosure of one's HIV status. The project aimed to use various psychometric tools to determine if these scores have a predictive value on late testing, treatment succes, quality of follow up, and disclosure of HIV to sex partners. The expected outcomes would be to be able to stratify patients using a behavioural risk score and allocate targeted ressources to improve the quality of care for the most at risk patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV Infected outpatient

Exclusion Criteria:

* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV Cohort
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2015-02; Primary Completion 2015-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
CD4 Count | 1 year after interview
  CD4 count at diagnosis and last recorded measure

SECONDARY OUTCOMES:
viral load | 1 year after interview
hiv disclosure to partner | at the time of interview
loss to follow up | one year after interview